CLINICAL TRIAL: NCT03874117
Title: Efficacy of Twice Weekly Hemodialysis in Patients With Residual Kidney Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Palo Alto Veterans Institute for Research (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Tammy Sirich, Principal Investigator, Palo Alto Veterans Institute for Research
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: SIT0003AGG; R01DK118426 (NIH)
Record Dates: First submitted 2019-03-10; First posted 2019-03-14 (Actual); Results first posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Hemodialysis; Kidney Failure, Chronic
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Twice Weekly Hemodialysis then Thrice Weekly Hemodialysis (Other): Twice weekly hemodialysis for 4 weeks, then thrice weekly hemodialysis for 4 weeks.
  Interventions: Other: Twice Weekly Hemodialysis then Thrice Weekly Hemodialysis
- Thrice Weekly Hemodialysis then Twice Weekly Hemodialysis (Other): Thrice weekly hemodialysis for 4 weeks, then twice weekly hemodialysis for 4 weeks.
  Interventions: Other: Thrice Weekly Hemodialysis then Twice Weekly Hemodialysis

INTERVENTIONS:
Other: Twice Weekly Hemodialysis then Thrice Weekly Hemodialysis — Twice weekly hemodialysis for 4 weeks, then thrice weekly hemodialysis for 4 weeks.
  Arms: Twice Weekly Hemodialysis then Thrice Weekly Hemodialysis
Other: Thrice Weekly Hemodialysis then Twice Weekly Hemodialysis — Thrice weekly hemodialysis for 4 weeks, then twice weekly hemodialysis for 4 weeks.
  Arms: Thrice Weekly Hemodialysis then Twice Weekly Hemodialysis

SUMMARY:
The study will determine the efficacy of twice weekly hemodialysis in patients with residual kidney function.

DETAILED DESCRIPTION:
Hemodialysis patients who have residual kidney function will undergo two 4-week study (twice weekly versus thrice weekly hemodialysis) using a cross-over design. Blood, urine, and dialysate samples will be collected at the end of each study period to determine adequacy of treatment and to assess uremic solute levels. Participants will complete quality of life questionnaires and cognitive paper tests.

ELIGIBILITY:
Inclusion Criteria:

* patients on hemodialysis who have residual kidney function with residual urea clearance (Kru) >2.5 mL/min.
* been on hemodialysis for at least 3 months.
* adherence to regular dialysis treatments.

Exclusion Criteria:

* inability to achieve adequate hemodialysis.
* planned revision of hemodialysis vascular access.
* hospitalized within the past 2 months.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2025-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tammy Sirich, MD, Principal Investigator — Stanford/VA Palo Alto Health Care System
Locations (3):
- United States (3):
  - VA Palo Alto Health Care System, Palo Alto, California
  - Santa Clara Valley Medical Center, San Jose, California
  - Satellite HealthCare, San Jose, California

REFERENCES:
- [Derived] Lee S, Pham NM, Montez-Rath ME, Bolanos CG, Bonde SS, Meyer TW, Sirich TL. Twice Weekly versus Thrice Weekly Hemodialysis-A Pilot Cross-Over Equivalence Trial. Clin J Am Soc Nephrol. 2024 Sep 1;19(9):1159-1168. doi: 10.2215/CJN.0000000000000507. Epub 2024 Jun 26. PMID 38922689

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 58 participants signed informed consent. 27 did not meet trial eligibility criteria during the run-in period and so were not randomized to the study periods. 31 participants were randomized to the study periods.
Groups:
- Twice Weekly Hemodialysis Then Thrice Weekly Hemodialysis: Participants will undergo hemodialysis twice per week for 4 weeks and then hemodialysis thrice per week for 4 weeks.
- Thrice Weekly Hemodialysis Then Twice Weekly Hemodialysis: Participants will undergo hemodialysis thrice per week for 4 weeks and then hemodialysis twice per week for 4 weeks.
Period: First Intervention (4 Weeks)
Arm/Group | Twice Weekly Hemodialysis Then Thrice Weekly Hemodialysis | Thrice Weekly Hemodialysis Then Twice Weekly Hemodialysis
Started | 15 | 16
Completed | 13 | 13
Not Completed | 2 | 3
Not completed — received kidney transplant | 1 | 0
Not completed — Coronavirus Disease 2019 (COVID-19) imposed restrictions on research | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — hospitalized for infection | 0 | 1
Period: Second Intervention (4 Weeks)
Arm/Group | Twice Weekly Hemodialysis Then Thrice Weekly Hemodialysis | Thrice Weekly Hemodialysis Then Twice Weekly Hemodialysis
Started | 13 | 13
Completed | 12 | 13
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Twice Weekly Hemodialysis Then Thrice Weekly Hemodialysis | Thrice Weekly Hemodialysis Then Twice Weekly Hemodialysis | Total
Number analyzed (Participants) | 15 | 16 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (11) | 59 (11) | 60 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 9 | 12 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 8 | 12
  Not Hispanic or Latino | 11 | 8 | 19
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 4 | 10
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 0 | 0 | 0
  White | 8 | 11 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Residual kidney urea clearance (Kru) [Mean (Standard Deviation); unit: mL/min] | 5.5 (2.1) | 4.2 (1.6) | 4.7 (1.9)

OUTCOME MEASURES:

1. Primary Outcome: QOL: Kidney Disease Quality of Life (KDQOL36)
Description: Kidney Disease Quality of Life: Health-related quality of life, with higher scores being better. Minimum is 0, maximum is 100.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Twice Weekly Hemodialysis: Participants who received twice weekly hemodialysis in either the first or last 4 weeks of the study.
- Thrice Weekly Hemodialysis: Participants who received thrice weekly hemodialysis in either the first or last 4 weeks of the study.
Arm/Group | Twice Weekly Hemodialysis | Thrice Weekly Hemodialysis
Number analyzed (Participants) | 26 | 25
score on a scale | 74 (17) | 72 (21)

2. Secondary Outcome: Solute Concentration
Description: Plasma concentration of p-cresol sulfate
Time Frame: 4 weeks
Measure: Mean (Inter-Quartile Range); unit: mg/dl
Arm/Group | Twice Weekly Hemodialysis | Thrice Weekly Hemodialysis
Number analyzed (Participants) | 26 | 25
mg/dl | 3.6 [2.5 to 4.6] | 3.6 [2.6 to 4.8]

3. Secondary Outcome: Symptom
Description: Dialysis Symptom Index: measures symptom burden on a scale of 0 to 150, with higher scores being worse.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Twice Weekly Hemodialysis | Thrice Weekly Hemodialysis
Number analyzed (Participants) | 26 | 25
score on a scale | 26 (26) | 32 (31)

4. Secondary Outcome: Trail B Making Test
Description: Cognitive test: The Trail B Making Test assesses working memory, cognitive flexibility, processing speed, and visual-motor tracking. There are numbers and letters on a page. The participant must connect the number to letter in order. For example, they would start at 1 and draw a line to A, then draw a line to 2, then draw a line to B, then draw a line to 3. The time is recorded in seconds.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Twice Weekly Hemodialysis | Thrice Weekly Hemodialysis
Number analyzed (Participants) | 26 | 25
seconds | 129 (73) | 125 (84)

5. Secondary Outcome: Digit Symbol Substitution Test
Description: Cognitive test: Digit Symbol Substitution Test, measured in number correct
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: number correct
Arm/Group | Twice Weekly Hemodialysis | Thrice Weekly Hemodialysis
Number analyzed (Participants) | 26 | 25
number correct | 51 (21) | 51 (20)

ADVERSE EVENTS:
Time Frame: 4 weeks for each intervention
Groups:
- Twice Weekly Hemodialysis: This intervention is when participants were on the twice weekly hemodialysis period for 4 weeks.
- Thrice Weekly Hemodialysis: This intervention is when participants were on the thrice weekly hemodialysis period for 4 weeks.
Arm/Group | Twice Weekly Hemodialysis | Thrice Weekly Hemodialysis
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/25
Other Adverse Events (participants affected / at risk) | 0/26 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2025-04-30): https://cdn.clinicaltrials.gov/large-docs/17/NCT03874117/Prot_000.pdf
  • Statistical Analysis Plan (2025-04-30): https://cdn.clinicaltrials.gov/large-docs/17/NCT03874117/SAP_001.pdf